CLINICAL TRIAL: NCT00677651
Title: Sex Differences in Gene Expression in Human Adipose Tissue
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: University of Maryland (Other)
Responsible Party: R. Jeffrey Chang, MD, University of California, San Diego
Other Study IDs: 070668
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Healthy; Obesity
Keywords: adipose; lean; obese; overweight; healthy
MeSH Terms: conditions — Obesity; Overweight | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Fat tissue from abdomen and buttock
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Five caucasian women
  Interventions: Procedure: Adipose Biopsy; Procedure: Blood sample; Radiation: CT Scan; Radiation: DEXA
- 2: Five caucasian men
  Interventions: Procedure: Adipose Biopsy; Procedure: Blood sample; Radiation: CT Scan; Radiation: DEXA

INTERVENTIONS:
Procedure: Adipose Biopsy — Adipose tissue will be sampled from the abdomen and buttock
Procedure: Blood sample — Blood will be sampled from an IV line
Radiation: CT Scan — Single image at the level of the liver
Radiation: DEXA — Whole body scan

SUMMARY:
This project was created to assess sex differences in adipose tissue gene expression in different locations in the body. The primary objectives are to understand:

1. The mechanisms of differential body fat distribution in men and women
2. How body fat distribution is affected by reproductive hormones
3. The mechanisms linking fat distribution to health risks such as diabetes

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women 20-35 years of age
* Lean (BMI less than 25)
* Obese (BMI 30-35)

Exclusion Criteria:

* Hormonal birth control
* Pregnancy
* Smokers
* History of diabetes, kidney, liver or thyroid disease
* History of cancer

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General Population
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Adipose and blood sampling | 1 year

SECONDARY OUTCOMES:
CT scan and DEXA scan | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Chang, M.D., Principal Investigator — UCSD
Locations (1):
- UCSD, La Jolla, California, United States